CLINICAL TRIAL: NCT03381612
Title: Prevalence of Female Circumcision Among Young Women in Beni-Suef, Egypt. A Cross-sectional Study
Brief Title: Prevalence of Female Circumcision Among Young Women in Beni-Suef, Egypt
Acronym: FC
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant Professor of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 14
Record Dates: First submitted 2017-12-08; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Woman Abuse
Keywords: Female circumcision, Young Women, Dysmenorrhea,Dysuria
MeSH Terms: conditions — Dysmenorrhea; Dysuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Female circumcision (FC) is a deeply-rooted practice in Egypt with deblitating physical and psychological consequences, however the previous two decades witnessed sincere efforts to counterfight this practice. The objective of this study is to investigate the prevalence of circumcision among young women (12-25 years) in Beni-Suef , Egypt.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on a total of 3353young women residing urban and rural quraters in Beni-Suef City. Data was collected usinga questionnaire that included information about the socio-demographic charcteristics of the women, their gynecological data, exposure to FC, and complaints associated with menses during the previous year.

ELIGIBILITY:
Inclusion Criteria:

* Young women aged 12 to 25 years living in Beni-Suef city of Egypt. the urban Metropolitan of Beni-Suef City was classified according to the socioeconomic level of its quarters to low, middle, and high levels. Out of each level, one quarter was selected randomly, by a card withdrawal, where households residing these quarters were chosen using a random start. For the rural villages surrounding the urban Metropolitan, three villages were selected randomly; one on the road to the North, one on the road to the West, and the last one on the road tothe South. Each village was clustered roughly into two sites; one to the East of the water channel and one to the West of the same water channel

Exclusion Criteria:

* Women from other places in Egypt.

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The urban Metropolitan of Beni-Suef City was classified according to the socioeconomic level of its quarters to low, middle, and high levels. Out of each level, one quarter was selected randomly, by a card withdrawal, where households residing these quarters were chosen using a random start. For the rural villages surrounding the urban Metropolitan, three villages were selected randomly; one on the road to the North, one on the road to the West, and the last one on the road to the South. Each village was clustered roughly into two sites; one to the East of the water channel and one to the West of the same water channel.
  In both urban and rural areas, a trained team of data collectors visited the selected households. Householders were informed briefly of the study and the residing women aged between 12 and 25 years were invited to participate and then interviewed.
Sampling Method: Probability Sample
Enrollment: 3353 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Gynecological manifestations measured by a questionnaire. | one year
  A questionnaire included questions about the manifestations associated with menses and average duration of dysmenorrhea during the previous year.

SECONDARY OUTCOMES:
social status measured by a questionnaire | one year
  A questionnaire included questions about age at menarche, social, educational and work status.

OTHER OUTCOMES:
working status measured by a questionnaire | One year
  For data collection, a questionnaireof two sections was prepared;the first section included socio-demographic data, social status, working status and educational level,age at menarche, menstrual cycle duration and flow days, in addition to exposure to circumcision. The second section includedquestions about the manifestations associated with menses and average duration of dysmenorrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burstyn L. Female circumcision comes to America. The Atlantic Monthly. 1995; pp 28-35.
- [Background] Moustafa T. Conflict and cooperation between the state and religious institutions in contemporary Egypt. International Journal of Middle East Studies 2000; 32:3-22.
- [Background] Sayed GH, Abd el-Aty MA, Fadel KA. The practice of female genital mutilation in upper Egypt. Int J Gynaecol Obstet. 1996 Dec;55(3):285-91. doi: 10.1016/s0020-7292(96)02753-1. PMID 9003955